CLINICAL TRIAL: NCT01589133
Title: A Multi-center Clinical Study for Assessment of the Consistency of the Results of Human Irregular Antibody Screening With Surgiscreen and Serascan Diana 3
Brief Title: Surgiscreen Registration
Status: Completed | Type: Observational
Sponsor: Johnson & Johnson Medical, China (Industry)
Responsible Party: Sponsor
Other Study IDs: OCD-201108
Record Dates: First submitted 2012-04-26; First posted 2012-05-01 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2012-04

CONDITIONS: Irregular Antibody Screening
Keywords: Irregular antibody screening

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma or Serum left after routine clinical testing.
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to assess the consistency of the results of irregular antibody screening with Surgiscreen （investigational reagent) and Serascan Diana 3 (control reagent), and the consistency of the results of irregular antibody screening with investigational reagent on serum and plasma from same patients.

ELIGIBILITY:
Inclusion Criteria:

* Serum or plasma samples left after routine clinical testing;
* Blood sample of the same day, or blood samples stored at 2-8°C for 3 days after collection, or serum or plasma samples stored at -20°C for those separated 3 days after collection.

Exclusion Criteria:

* Samples with severe hemolysis, jaundice or chyle-like samples;
* Small sample size insufficient for completing the testing;
* Samples not collected and processed upon the requirements of the instructions.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who need transfusion therapy in investigator sites.
Sampling Method: Non-Probability Sample
Enrollment: 3109 (Actual)
Dates: Start 2012-05; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
The consistency of the results of irregular antibody screening of investigational reagent and control reagent. | baseline
  The positive coincidence rate, the negative coincidence rate and the overall coincidence rate, as well as their respective 95% confidence interval of the irregular antibody screening results of two reagents.

SECONDARY OUTCOMES:
The consistency of the results of irregular antibody screening with investigational reagent on different types of samples (serum and plasma). | baseline
  The positive coincidence rate, the negative coincidence rate and the overall coincidence rate, as well as their respective 95% confidence interval of the irregular antibody screening results of investigational reagent on serum and plasma from same patient.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Cancer Institute & Hospital, Chinese Academy of Medical Science, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality
  - Shanghai Blood Center, Shanghai, Shanghai Municipality